CLINICAL TRIAL: NCT00851526
Title: Coronary Bifurcation Stenting (COBIS) Registry in South Korea
Acronym: COBIS
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Other Study IDs: 2007-04-042
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Bifurcation Lesion
Keywords: Coronary bifurcation lesion; Drug-eluting stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Coronary bifurcation lesion

SUMMARY:
The COBIS registry is multi-center, real-world registry of drug-eluting stenting in coronary bifurcation lesions in South Korea.

The aim of the study was to find out the current status of bifurcation drug-eluting stenting and determine the prognostic factors for long-term outcome in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Any type of de novo bifurcation lesion with a parent vessel >= 2.5 mm and side branch>= 2.0 mm by visual estimation
* Treated with drug-eluting stent

Exclusion Criteria:

* Cardiogenic Shock
* ST elevation MI within 48hours
* Expected survival less than 1 year
* Left main bifurcation
* Allergy to the antiplatelets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary bifurcation lesion treated with drug-eluting stents
Sampling Method: Probability Sample
Enrollment: 1919 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Incidence of the composite outcome of all-cause death, MI, or any PCI/CABG | 3 years

SECONDARY OUTCOMES:
Incidence of stent thrombosis, and periprocedural MI | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song PS, Song YB, Yang JH, Hahn JY, Choi SH, Choi JH, Koo BK, Seung KB, Park SJ, Gwon HC. The impact of side branch predilatation on procedural and long-term clinical outcomes in coronary bifurcation lesions treated by the provisional approach. Rev Esp Cardiol (Engl Ed). 2014 Oct;67(10):804-12. doi: 10.1016/j.rec.2014.01.032. Epub 2014 Jul 10. PMID 25262126
- [Derived] Chung S, Her SH, Song PS, Song YB, Hahn JY, Choi JH, Lee SH, Jang Y, Yoon JH, Tahk SJ, Park SJ, Choi SH, Seung KB, Gwon HC. Trans-radial versus trans-femoral intervention for the treatment of coronary bifurcations: results from Coronary Bifurcation Stenting Registry. J Korean Med Sci. 2013 Mar;28(3):388-95. doi: 10.3346/jkms.2013.28.3.388. Epub 2013 Mar 4. PMID 23486858
- [Derived] Song PS, Song YB, Yang JH, Kang GH, Hahn JY, Choi SH, Choi JH, Lee SH, Jang Y, Yoon JH, Tahk SJ, Seung KB, Park SJ, Gwon HC. Periprocedural myocardial infarction is not associated with an increased risk of long-term cardiac mortality after coronary bifurcation stenting. Int J Cardiol. 2013 Aug 20;167(4):1251-6. doi: 10.1016/j.ijcard.2012.03.146. Epub 2012 Apr 9. PMID 22494861
- [Derived] Gwon HC, Hahn JY, Koo BK, Song YB, Choi SH, Choi JH, Lee SH, Jeong MH, Kim HS, Seong IW, Yang JY, Rha SW, Jang Y, Yoon JH, Tahk SJ, Seung KB, Park SJ. Final kissing ballooning and long-term clinical outcomes in coronary bifurcation lesions treated with 1-stent technique: results from the COBIS registry. Heart. 2012 Feb;98(3):225-31. doi: 10.1136/heartjnl-2011-300322. Epub 2011 Sep 20. PMID 21933939
- [Derived] Gwon HC, Choi SH, Song YB, Hahn JY, Jeong MH, Seong IW, Kim HS, Rha SW, Yang JY, Yoon JH, Tahk SJ, Seung KB, Jang Y, Park SJ. Long-term clinical results and predictors of adverse outcomes after drug-eluting stent implantation for bifurcation lesions in a real-world practice: the COBIS (Coronary Bifurcation Stenting) registry. Circ J. 2010 Nov;74(11):2322-8. doi: 10.1253/circj.cj-10-0352. Epub 2010 Sep 28. PMID 20890049
- [Derived] Song YB, Hahn JY, Choi SH, Choi JH, Lee SH, Jeong MH, Kim HS, Seong IW, Yang JY, Rha SW, Jang Y, Yoon JH, Tahk SJ, Seung KB, Park SJ, Gwon HC. Sirolimus- versus paclitaxel-eluting stents for the treatment of coronary bifurcations results: from the COBIS (Coronary Bifurcation Stenting) Registry. J Am Coll Cardiol. 2010 Apr 20;55(16):1743-50. doi: 10.1016/j.jacc.2010.02.008. PMID 20394879